CLINICAL TRIAL: NCT05051319
Title: Investigation of Factors Associated With Cognitive Status in the Elderly
Brief Title: Factors Associated With Cognitive Status in the Elderly
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, Principal Investıgator, Pamukkale University
Other Study IDs: 60116787-020/16528
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Elderly

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly participants living at home: Participants over the age of 65, living at home, not having mental and communication problems that would prevent the evaluations, and volunteering to participate in the study. The sociodemographic information of the participants such as gender, duration of education, living environment and people with whom they live were recorded. In addition, information about the medical condition of geriatric individuals, such as body mass indexes and the number of drugs used, was also recorded in the form. In order to evaluate the cognitive status of the participants, the Standardized or Standardized Mini-Mental Test for the Uneducated was used according to their educational status. The Center for Disease Control Health-Related Quality of Life-4 Scale (CDC HRQoL-4) was used to assess quality of life, and the Geriatric Depression Scale was used to assess emotional status. In addition, the presence of pain and pain levels according to body regions were determined with a 6-point Likert-type scale.

SUMMARY:
The aim of this study was to investigate the factors related to cognitive status in elderly individuals living in the community. A total of 841 elderly (female: 422, male: 419) living in the community were included in this cross-sectional study. The sociodemographic information of the elderly was recorded. In addition, cognitive status, quality of life, depression and musculoskeletal pain were questioned. The classification and regression tree analysis was used to identify factors associated with cognitive status. Age, depression, quality of life, neck pain, and headache were determinative on the cognitive status of the elderly. Knowing the factors related to cognitive status in elderly individuals living in the community is very important in terms of early diagnosis of factors that may affect the quality of life of these individuals.

DETAILED DESCRIPTION:
Aim: The aim of this study was to investigate the factors related to cognitive status in elderly individuals living in the community.

Methods: A total of 841 elderly (female: 422, male: 419) living in the community were included in this cross-sectional study. The sociodemographic information of the elderly was recorded. In addition, cognitive status, quality of life, depression and musculoskeletal pain were questioned. The classification and regression tree analysis was used to identify factors associated with cognitive status.

ELIGIBILITY:
Inclusion Criteria:

* Participants over the age of 65,
* Living at home,
* Not having mental and communication problems that would prevent the evaluations,
* Volunteering to participate in the study.

Exclusion Criteria:

* Central nervous system diseases affecting cognitive functions.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly participants was included the study residing in the city center of Denizli, living at home, having no communication and mental disability problems that would affect the evaluations, and giving informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Center for Disease Control and Prevention Health-Related Quality of Life-4 Scale | Two years
  The quality of life of the elderly participants was evaluated with the first question of the CDC HRQOL-4 scale. The Turkish validity-reliability study of the scale is a short and understandable scale used to evaluate the quality of life. This scale consists of 4 questions evaluating the general health of the participants, their physical and mental health in the last 30 days, and how activities such as self-care, work, school, and hobbies have been affected by their physical or mental problems in the last 30 days. In question 1, general health was defined as excellent, very good, good, fair, and poor. In the 2nd, 3rd, and 4th questions, the number of days in the last 30 days when the participant felt unwell physically and mentally, and the number of days the person could not perform his daily activities due to physical and/or mental problems are recorded.
Standardized Mini-Mental Test | Two years
  Standardized Mini-Mental Test was applied to determine the cognitive levels of the participants. For the illiterate elderly, SMMT, which is used for the uneducated, was applied in our study. In this test, orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points) were collected under 5 main headings. It consists of 11 items and is evaluated over a total of 30 points. Results; 27-30 points are within normal limits, 24-27 points are mild cognitive impairment, below 24 points are considered severe cognitive impairment. The Turkish validity and reliability study of the questionnaire was conducted in 2002.
Geriatric Depression Scale | Two years
  The scale was prepared for the geriatric individuals to easily mark and answer "yes" or "no". It consists of 30 questions. In the scoring of the scale, 1 point is given for each response in favor of depression and 0 point is given for the other answer, and the result is accepted as the depression score. Scoring of the scale was made as "no depression" with 0-10 points, "possible depression" with 11 points, and "definite depression" with 14 and above points. When 14 is taken as the threshold value for Geriatric Depression Scale scores, its specificity approaches 100%. A validity and reliability study of the Geriatric Depression Scale was conducted in the Turkish elderly population.
Assessment of Pain | Two years
  The chronic pain status in 10 different body regions of the individuals were assessed in the study. The presence of pain (present or absent) and severity of pain in geriatric individuals were evaluated with a 6-point Likert-type scale (0=no pain, 1=mild, 2=moderate, 3=severe, 4=very severe, 5=unbearable). This pain scale was preferred in order to make it easier for geriatric individuals to understand the severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Güzin Kara, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kınıklı/Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Arnim CAF, Bartsch T, Jacobs AH, Holbrook J, Bergmann P, Zieschang T, Polidori MC, Dodel R. Diagnosis and treatment of cognitive impairment. Z Gerontol Geriatr. 2019 Jul;52(4):309-315. doi: 10.1007/s00391-019-01560-0. Epub 2019 Jun 3. PMID 31161337
- [Result] Li CL, Hsu HC. Cognitive function and associated factors among older people in Taiwan: age and sex differences. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):196-200. doi: 10.1016/j.archger.2014.10.007. Epub 2014 Oct 17. PMID 25456889
- [Result] Kloszewska M, Lyszczarz B, Kedziora-Kornatowska K. Sociodemographic and Health-Related Factors Associated with Severity of Cognitive Impairment in Elderly Patients Hospital-ized in a Geriatric Clinic. Brain Sci. 2021 Jan 29;11(2):170. doi: 10.3390/brainsci11020170. PMID 33572984